CLINICAL TRIAL: NCT02270125
Title: The Role of Nanoparticles in Inflammatory Changes of the Nasal Mucosa
Brief Title: Nanoparticles in Nasal Mucosa
Status: Completed | Type: Observational
Sponsor: University Hospital Ostrava (Other)
Collaborators: VSB - Technical University of Ostrava (Unknown)
Responsible Party: Sponsor
Other Study IDs: FNO-ENT-Nanoparticles; 2 RVO-FNOs/2013 (Other Grant/Funding Number: Ministry of Health of the Czech Republic)
Record Dates: First submitted 2014-10-13; First posted 2014-10-21 (Estimated); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hypertrophic Rhinosinusitis; Chronic Polypous Rhinosinusitis
Keywords: nasal mucosa; chronic hypertrophic rhinosinusitis; mucotomy; nanoparticles; scanning electron microscopy; Raman microspectroscopy; nasal polyposis
MeSH Terms: conditions — Nasal Polyps

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — nasal mucosa of the inferior nasal turbinate obtained by mucotomy in adult pacients nasal mucosa of the inferior nasal turbinate obtained by mucotomy in stillborn children
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Adult patients with chronic rhino sinusitis: Group of adult patients indicated for mucotomy due to chronic hypertrophic rhinosinusitis, with or without polyposis
  Interventions: Procedure: Mucotomy
- Stillborn children: Control group of stillborn children whose nasal mucosa was not exposed to airborne particles
  Interventions: Procedure: Mucotomy

INTERVENTIONS:
Procedure: Mucotomy — Surgical removal of hypertrophic mucosa of the inferior nasal turbinate by cold-steel instruments under endoscopic control, under general anaesthesia
  Other Names: turbinoplasty

SUMMARY:
The aim of this prospective study is to evaluate presence and quantity of nano-sized particles and interindividual differences in their distribution and elemental composition in human nasal mucosa obtained by mucotomy in patients diagnosed with chronic hypertrophic rhinosinusitis and to compare the obtained results with control specimen obtained from stillborn children.

DETAILED DESCRIPTION:
Samples of nasal mucosa are obtained by mucotomy in general anesthaesia from adult patients with chronic hypertrophic rhinosinusitis. Each tissue sample is divided into 4 parts based on the distance from the nostrils and is dehydrated, thinly sliced and mounted on glass slides. Then the tissue is analyzed with scanning electron microscopy (SEM) and Raman microspectroscopy (RMS) to detect solid particles and characterize the morphology and compositions of the detected particles. A novel method of quantification of distribution of the particles has been designed and used to evaluate interindividual differences in distribution of the particles. History of employment is obtained from the patients and the data are compared with the findings in the tissue samples.

The data acquired from the group of adult patients are compared with the results obtained from a group of control specimen of nasal mucosa harvested from stillborn children. It is presumed that no nano particles will be present in the stillborn children specimen since the mucosa was not exposed to airborne particles.

ELIGIBILITY:
Inclusion Criteria:

* chronic hypertrophic rhihosinusitis without polyposis non responsive to conservative treatment for at least six months
* chronic hypertrophic rhihosinusitis with polyposis non responsive to conservative treatment for at least six months
* age between 19 and 64 years of age
* signed informed consent of the patient
* stillborn children born after 28th week of gestation

Exclusion Criteria:

- non-signing of the informed consent

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adult patients with chronic hypertrophic rhinosinusitis, with or without polyposis Stillborn children
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2013-09; Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Detection and characterisation of nano particles | 36 months
  Morphology characterization and elemental composition of the particles found in the nasal mucosa assessed with SEM (Quanta FEG 450, FEI) with X-ray microanalysis APOLLO X (EDAX) and SEM Philips XL 30 operating at 30 keV.

SECONDARY OUTCOMES:
The presence of nano particles in the nasal mucosa obtained from stillborn children | 36 months
  Confirmation of the presence of nano particle in the nasal mucosa obtained from stillborn children (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Lenka Čábalová, MD, Principal Investigator — University Hospital Ostrava, Medical Faculty of the Ostrava University
Locations (2):
- Czechia (2):
  - Nanotechnology Centre, VSB-Technical University Ostrava, Ostrava, Czech Republic
  - University Hospital Ostrava, Ostrava, Czech Republic

REFERENCES:
- [Background] Zelenik K, Kukutschova J, Dvorackova J, Bielnikova H, Peikertova P, Cabalova L, Kominek P. Possible role of nano-sized particles in chronic tonsillitis and tonsillar carcinoma: a pilot study. Eur Arch Otorhinolaryngol. 2013 Feb;270(2):705-9. doi: 10.1007/s00405-012-2069-5. Epub 2012 Jun 8. PMID 22678622
- [Background] Dvorackova J, Bielnikova H, Kukutschova J, Peikertova P, Filip P, Zelenik K, Kominek P, Uvirova M, Pradna J, Cermakova Z, Dvoracek I. Detection of nano- and micro-sized particles in routine biopsy material - pilot study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2015 Mar;159(1):87-92. doi: 10.5507/bp.2012.104. Epub 2012 Dec 10. PMID 23235723
- [Background] Oberdorster G, Oberdorster E, Oberdorster J. Nanotoxicology: an emerging discipline evolving from studies of ultrafine particles. Environ Health Perspect. 2005 Jul;113(7):823-39. doi: 10.1289/ehp.7339. PMID 16002369